CLINICAL TRIAL: NCT00337428
Title: An Open-Label, Randomized, Multicenter Study of the Safety, Tolerability, and Immunogenicity of Gardasil (V501) Given Concomitantly With REPEVAX™ in Healthy Adolescents 11-17 Years of Age
Brief Title: Concomitant Use of Gardasil (V501, Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine) With Combined Diptheria, Tetanus, Pertussis and Poliomyelitis Vaccine in Adolescents (V501-024)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V501-024; 2005_093
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: Neoplasms, Glandular and Epithelial; Diphtheria; Tetanus; Whooping Cough; Poliomyelitis
MeSH Terms: conditions — Neoplasms, Glandular and Epithelial; Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

ARMS (4):
- Group 1 (Experimental): Concomitant/CMF
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Current Manufacturing Facility (CMF); Biological: Comparator: REPEVAX™ (Concomitant)
- Group 2 (Experimental): Non-Concomitant/CMF
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Current Manufacturing Facility (CMF); Biological: Comparator: REPEVAX™ (Non-Concomitant)
- Group 3 (Experimental): Concomitant/FMF
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Future Manufacturing Facility (FMF); Biological: Comparator: REPEVAX™ (Concomitant)
- Group 4 (Experimental): Non-Concomitant/FMF
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Future Manufacturing Facility (FMF); Biological: Comparator: REPEVAX™ (Non-Concomitant)

INTERVENTIONS:
Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Current Manufacturing Facility (CMF) — GARDASIL™ (quadrivalent human papillomavirus [types 6, 11, 16, 18] virus-like particle [VLP] vaccine, referred to as qHPV vaccine) made at the current manufacturing facility was administered as 0.5-mL intramuscular dose at Day 1, Month 2, and Month 6.
  Arms: Group 1; Group 2
Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) Vaccine from Future Manufacturing Facility (FMF) — GARDASIL™ (quadrivalent human papillomavirus [types 6, 11, 16, 18] virus-like particle [VLP] vaccine, referred to as qHPV vaccine) made at the future manufacturing facility was administered as 0.5-mL intramuscular dose at Day 1, Month 2, and Month 6.
  Arms: Group 3; Group 4
Biological: Comparator: REPEVAX™ (Concomitant) — REPEVAX™ (diphtheria, tetanus, pertussis [acellular, component] and poliomyelitis [inactivated] vaccine, Sanofi Pasteur, Swiftwater, PA U.S.A) was administered as a single 0.5-mL intramuscular dose at Day 1 in a limb opposite that of quadrivalent HPV injection.
  Arms: Group 1; Group 3
Biological: Comparator: REPEVAX™ (Non-Concomitant) — REPEVAX™ (diphtheria, tetanus, pertussis [acellular, component] and poliomyelitis [inactivated] vaccine, Sanofi Pasteur, Swiftwater, PA U.S.A) was administered as a single 0.5-mL intramuscular dose at Month 1 in a limb opposite that of quadrivalent HPV injection.
  Arms: Group 2; Group 4

SUMMARY:
Data from this study are expected to demonstrate that Gardasil (V501, Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine), when administered concomitantly with a combined diphtheria, tetanus, pertussis, and poliomyelitis vaccine in adolescents remains immunogenic and well-tolerated and it does not impair the immunogenicity of the concomitant vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy boys or girls, 11-17 years of age
* Must be a virgin with no intention of becoming sexually active during the study period
* Must have been properly vaccinated against diphtheria, tetanus, pertussis and polio

Exclusion Criteria:

* Must not have received a vaccine against diphtheria, tetanus, pertussis and polio in the past 5 years
* Must not have received any prior human papillomavirus (HPV) vaccine

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 843 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Vesikari T, Van Damme P, Lindblad N, Pfletschinger U, Radley D, Ryan D, Vuocolo S, Haupt RM, Guris D. An open-label, randomized, multicenter study of the safety, tolerability, and immunogenicity of quadrivalent human papillomavirus (types 6/11/16/18) vaccine given concomitantly with diphtheria, tetanus, pertussis, and poliomyelitis vaccine in healthy adolescents 11 to 17 years of age. Pediatr Infect Dis J. 2010 Apr;29(4):314-8. doi: 10.1097/INF.0b013e3181c177fb. PMID 19952980

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled healthy participants, 11-17 years old, with 0 lifetime sexual partners, vaccinated against diphtheria, tetanus, pertussis and polio but had not received the vaccine in the past 5 years or any prior human papillomavirus (HPV) vaccine. Additional inclusion and exclusion criteria applied.
Groups:
- qHPV Vaccine + REPEVAX™ (Concomitant): Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) vaccine and REPEVAX™ administered on Day 1 at different injection sites.
- qHPV Vaccine + REPEVAX™ (Non-Concomitant): Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant (qHPV) vaccine administered on Day 1 followed by REPEVAX™ administered at Month 1.
Period: Overall Study
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Started | 419 | 424
Completed | 415 | 421
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Time | 1 | 1
Not completed — Unwilling to Continue | 1 | 0
Not completed — Anorexia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant) | Total
Number analyzed (Participants) | 419 | 424 | 843
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (1.5) | 12.1 (1.5) | 12.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 288 | 583
  Male | 124 | 136 | 260
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 4
  Black | 3 | 3 | 6
  Multi-racial | 2 | 3 | 5
  White | 413 | 415 | 828

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 6 at Month 7 (4 Weeks Postdose 3)
Description: Serum antibodies to HPV Type 6 were measured with a Competitive Luminex Immunoassay. Titers were reported in milli Merck Units (mMU)/milliliter (mL). GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs for each HPV type using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: Per-protocol population: participants must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data.
Measure: Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 367 | 376
milliMerck units/mL | 1151.3 [1007.5 to 1315.7] | 1244.9 [1092.4 to 1418.6]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

2. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 11 at Month 7 (4 Weeks Postdose 3)
Description: Serum antibodies to HPV Type 11 were measured with a Competitive Luminex Immunoassay. Titers were reported in milli Merck Units (mMU)/milliliter (mL). GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs for each HPV type using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 367 | 376
milliMerck units/mL | 1338.3 [1209.0 to 1481.4] | 1460.7 [1322.4 to 1613.3]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

3. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 16 at Month 7 (4 Weeks Postdose 3)
Description: Serum antibodies to HPV Type 16 were measured with a Competitive Luminex Immunoassay. Titers were reported in milli Merck Units (mMU)/milliliter (mL). GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs for each HPV type using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 370 | 378
milliMerck units/mL | 5835.7 [5195.7 to 6554.6] | 6508.1 [5810.3 to 7289.6]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

4. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 18 at Month 7 (4 Weeks Postdose 3)
Description: Serum antibodies to HPV Type 18 were measured with a Competitive Luminex Immunoassay. Titers were reported in milli Merck Units (mMU)/milliliter (mL). GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs for each HPV type using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliMerck units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 372 | 378
milliMerck units/mL | 1096.0 [958.8 to 1252.8] | 1308.8 [1148.1 to 1491.9]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

5. Primary Outcome: Number of Participants Who Seroconverted for HPV Type 6 (HPV 6 ≥20 mMU/mL) by Month 7 (4 Weeks Postdose 3)
Description: Seroconversion to HPV Type 6 was defined as changing serostatus from seronegative to seropositive as measured by GMT. The cutoff value for HPV seropositivity was ≥20 mMU/mL. Seroconversion of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) was compared to seroconversion of participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared seroconversion for each HPV type using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 367 | 376
participants | 367 | 375
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

6. Primary Outcome: Number of Participants Who Seroconverted for HPV Type 11 (HPV 11 ≥16 mMU/mL) by Month 7 (4 Weeks Postdose 3)
Description: Seroconversion to HPV Type 11 was defined as changing serostatus from seronegative to seropositive as measured by GMT. The cutoff value for HPV seropositivity was ≥16 mMU/mL. Seroconversion of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) was compared to seroconversion of participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared seroconversion for each HPV type using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 367 | 376
participants | 367 | 376
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

7. Primary Outcome: Number of Participants Who Seroconverted for HPV Type 16 (HPV 16 ≥20 mMU/mL) by Month 7 (4 Weeks Postdose 3)
Description: Seroconversion to HPV Type 16 was defined as changing serostatus from seronegative to seropositive as measured by GMT. The cutoff value for HPV seropositivity was ≥20 mMU/mL. Seroconversion of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) was compared to seroconversion of participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared seroconversion for each HPV type using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 370 | 378
participants | 370 | 378
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

8. Primary Outcome: Number of Participants Who Seroconverted for HPV Type 18 (HPV 18 ≥24 mMU/mL) by Month 7 (4 Weeks Postdose 3)
Description: Seroconversion to HPV Type 18 was defined as changing serostatus from seronegative to seropositive as measured by GMT. The cutoff value for HPV seropositivity was ≥24 mMU/mL. Seroconversion of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) was compared to seroconversion of participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared seroconversion for each HPV type using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 7 Months (4 Weeks Postdose 3)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 372 | 378
participants | 372 | 378
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

9. Primary Outcome: Number of Participants Who Achieved Acceptable Levels of Titers to Diphtheria (Diphtheria ≥0.1 IU/mL) One Month Post-vaccination With REPEVAX™
Description: Diphtheria antitoxin titers were measured using a neutralization assay in Vero cell culture that compares the antitoxin level in the serum of participants with the World Health Organization International Standard for Diphtheria Antitoxin. An acceptable level of response was defined as ≥0.1 International Units (IU)/milliliter (mL). Response levels of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared response levels using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 380 | 380
participants | 380 | 379
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

10. Primary Outcome: Number of Participants Who Achieved Acceptable Levels of Titers to Tetanus (Tetanus ≥0.1 IU/mL) One Month Post-vaccination With REPEVAX™
Description: Tetanus antitoxin titers were measured using an indirect, non-competitive enzyme immunoassay (EIA) that compares the antitoxin level in the serum of participants with the World Health Organization International Standard for Tetanus Immunoglobulin. An acceptable level of response was defined as ≥0.1 International Units (IU)/milliliter (mL). Response levels of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared response levels using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 381 | 380
participants | 381 | 380
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

11. Primary Outcome: Number of Participants Who Achieved Acceptable Levels of Titers to Poliovirus Type 1 (Poliovirus Type 1 ≥1:8) One Month Postvaccination With REPEVAX™
Description: Poliovirus antibody was measured using a poliovirus neutralization assay that assesses the ability of serial dilutions of participant sera to neutralize known amounts of type-specific Sabin poliovirus strains (Types 1, 2, and 3). An acceptable level of response was defined as participants who achieve detectable serum neutralizing antibodies at a ≥1:8 dilution of sera. The response of participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) was compared to participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared response levels using methods developed by Miettinen and Nurminen adjusting for manufacturing facility for qHPV vaccine.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 367 | 377
participants | 367 | 376
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

12. Primary Outcome: Number of Participants Who Achieved Acceptable Levels of Titers to Poliovirus Type 2 (Poliovirus Type 2 ≥1:8) One Month Postvaccination With REPEVAX™
Description: as for outcome 11
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 369 | 377
participants | 369 | 376
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

13. Primary Outcome: Number of Participants Who Achieved Acceptable Levels of Titers to Poliovirus Type 3 (Poliovirus Type 3 ≥1:8) One Month Postvaccination With REPEVAX™
Description: as for outcome 11
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: participants
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 361 | 375
participants | 360 | 375
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions; Stat Med 1985;4:213-26

14. Primary Outcome: Geometric Mean Titers (GMTs) For Pertussis (Anti-PT) One Month Postvaccination With REPEVAX™
Description: Serum antibodies to Pertussis Toxoid Antibody (anti-PT) were measured with an enzyme-linked immunosorbent assay (ELISA). Titers were reported in ELISA units/mL (ELU/mL) and the lower limit of quantitation for the assay was 5.0 ELU/mL. GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 381 | 378
ELISA units/mL | 38.1 [33.2 to 43.7] | 35.7 [31.1 to 40.9]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

15. Primary Outcome: Geometric Mean Titers (GMTs) For Pertussis (Anti-FHA) One Month Postvaccination With REPEVAX™
Description: Serum antibodies to Pertussis Filamentous Haemagglutin Antibody (anti-FHA) were measured with an ELISA. Titers were reported in ELU/mL and the lower limit of quantitation for the assay was 3.0 ELU/mL. GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 382 | 381
ELISA units/mL | 140.3 [127.5 to 154.4] | 140.7 [127.9 to 154.7]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

16. Primary Outcome: Geometric Mean Titers (GMTs) For Pertussis (Anti-PRN) One Month Postvaccination With REPEVAX™
Description: Serum antibodies to Pertussis Pertactin (anti-PRN) were measured with an ELISA. Titers were reported in ELU/mL and the lower limit of quantitation for the assay was 5.0 ELU/mL. GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 382 | 381
ELISA units/mL | 504.1 [442.7 to 574.0] | 552.8 [485.9 to 629.1]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

17. Primary Outcome: Geometric Mean Titers (GMTs) For Pertussis (Anti-FIM) One Month Postvaccination With REPEVAX™
Description: Serum antibodies to Pertussis Fimbrial Agglutinogens Antibody (anti-FIM) were measured with an ELISA. Titers were reported in ELU/mL and the lower limit of quantitation for the assay was 5.0 ELU/mL. GMTs from participants who received qHPV vaccine and REPEVAX™ together at Day 1 (concomitant) were compared to GMTs from participants who received qHPV vaccine at Day 1 followed by REPEVAX™ 1 month later (non-concomitant). An analysis of non-inferiority compared GMTs for each HPV Type using an ANOVA model with a response of log individual titers and fixed effects for treatment group, manufacturing facility, study site, and the treatment-by-site interaction.
Time Frame: Up to 1 Month (1 Month Postdose 1)
Population: Per-protocol population: participants must have no major protocol violations and must have post-vaccination data.
Measure: Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Number analyzed (Participants) | 381 | 381
ELISA units/mL | 561.2 [478.9 to 657.7] | 506.4 [432.5 to 592.8]
Statistical Analysis 1: Comparison: qHPV Vaccine + REPEVAX™ (Concomitant) vs qHPV Vaccine + REPEVAX™ (Non-Concomitant); Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 1 until Month 7.
Description: AEs were collected on participants who received ≥1 dose of study vaccine (qHPV or Repevax). Fevers and injection-site AEs were reported for Days 1-5 and all other AEs for Days 1-15. Injection-site AEs are reported separately for those associated with qHPV (AE term-qHPV) and those that are associated with Repevax (AE term-Repevax).
Arm/Group | qHPV Vaccine + REPEVAX™ (Concomitant) | qHPV Vaccine + REPEVAX™ (Non-Concomitant)
Serious Adverse Events (participants affected / at risk) | 1/420 | 3/423
Other Adverse Events (participants affected / at risk) | 405/420 | 406/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine + REPEVAX™ (Concomitant) (N=420) | qHPV Vaccine + REPEVAX™ (Non-Concomitant) (N=423)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine + REPEVAX™ (Concomitant) (N=420) | qHPV Vaccine + REPEVAX™ (Non-Concomitant) (N=423)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 20 (26) | 12 (16)
Abdominal pain upper (Gastrointestinal disorders) | 14 (15) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 18 (21)
Nausea (Gastrointestinal disorders) | 21 (27) | 19 (21)
Vomiting (Gastrointestinal disorders) | 11 (11) | 11 (13)
Fatigue (General disorders) | 13 (13) | 8 (8)
Malaise (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 50 (53) | 55 (60)
Injection site bruising-qHPV (General disorders) | 6 (6) | 5 (5)
Injection site erythema-qHPV (General disorders) | 77 (98) | 63 (85)
Injection site haematoma-qHPV (General disorders) | 5 (5) | 7 (8)
Injection site induration-qHPV (General disorders) | 4 (4) | 5 (5)
Injection site pain-qHPV (General disorders) | 335 (641) | 304 (630)
Injection site pruritus-qHPV (General disorders) | 8 (8) | 11 (11)
Injection site swelling-qHPV (General disorders) | 89 (131) | 90 (119)
Injection site bruising-Repevax (General disorders) | 4 (4) | 2 (2)
Injection site erythema-Repevax (General disorders) | 77 (77) | 79 (80)
Injection site haematoma-Repevax (General disorders) | 3 (3) | 4 (4)
Injection site induration-Repevax (General disorders) | 3 (3) | 3 (3)
Injection site irritation-Repevax (General disorders) | 4 (4) | 5 (5)
Injection site pain-Repevax (General disorders) | 350 (383) | 346 (373)
Injection site pruritus-Repevax (General disorders) | 4 (4) | 7 (7)
Injection site swelling-Repevax (General disorders) | 130 (132) | 131 (132)
Injection site warmth-Repevax (General disorders) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 11 (12) | 10 (13)
Nasopharyngitis (Infections and infestations) | 25 (25) | 28 (29)
Pharyngitis (Infections and infestations) | 6 (6) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7)
Rhinitis (Infections and infestations) | 19 (21) | 20 (23)
Sinusitis (Infections and infestations) | 6 (6) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 21 (23) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 6 (8)
Dizziness (Nervous system disorders) | 14 (15) | 10 (11)
Headache (Nervous system disorders) | 132 (193) | 112 (168)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (4) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 11 (11)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 24 (29)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2)
Axillary pain (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 3 (3) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 3 (3) | 2 (2)
Local swelling (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (2) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 10 (11) | 7 (9)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 2 (4)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Listless (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Injection site irritation-qHPV (General disorders) | 1 (2) | 2 (2)
Injection site warmth-qHPV (General disorders) | 1 (1) | 2 (3)
Injection site anaesthesia-Repevax (General disorders) | 1 (1) | 1 (1)
Injection site discolouration-qHPV (General disorders) | 1 (1) | 1 (1)
Injection site discolouration-Repevax (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage-qHPV (General disorders) | 3 (3) | 4 (4)
Injection site haemorrhage-Repevax (General disorders) | 0 (0) | 1 (1)
Injection site mass-Repevax (General disorders) | 1 (1) | 0 (0)
Injection site movement impairment-qHPV (General disorders) | 1 (2) | 3 (5)
Injection site movement impairment-Repevax (General disorders) | 3 (3) | 3 (3)
Injection site nodule-qHPV (General disorders) | 1 (1) | 0 (0)
Injection site nodule-Repevax (General disorders) | 1 (1) | 0 (0)
Injection site papule-Repevax (General disorders) | 0 (0) | 1 (1)
Injection site rash-Repevax (General disorders) | 1 (1) | 0 (0)
Injection site reaction-qHPV (General disorders) | 1 (1) | 1 (1)
Injection site reaction-Repevax (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Safety results have been previously reported in the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.